CLINICAL TRIAL: NCT04129645
Title: Prospective Observational Study for Assessment of the Efficacy and Safety of Allium Ureteral Stent Long-term Indwelling in the Treatment of Ureteral Stricture
Brief Title: Safety and Efficacy of URS Stents in the Treatment of Ureteral Stricture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Huhao, Primary Investigator, Peking University People's Hospital
Other Study IDs: URO-01
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Ureteral Stricture
Keywords: Ureteral; ureteral stent; ureteral stricture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: URS — URS is a permanent ureteral stent made of nitinol and covered by a polymer, that is indicated to open strictures in the ureter.
  Study patients who has strictures in the ureter, will be implanted with the URS for long term opening of the stricture.

SUMMARY:
A prospective observational study aimed to assess the efficacy and safety of Allium ureteral stent long-term indwelling in the treatment of ureteral stricture.

ELIGIBILITY:
Inclusion Criteria:

1. Benign diseases: UPJ, ischemic injury caused by surgical separation, endoscopic surgery injury, heat injury by laser lithotripsy, infection (chronic inflammation, tuberculosis), peri-ureteral fibrosis caused by endometriosis, ureteral anastomotic stenosis after renal transplantation, ureteral fistula, multiple polyps;
2. Malignant diseases: ureteral anastomotic stricture after urinary diversion, stricture caused by compression of abdominal and/or pelvic tumors, stricture caused by urinary tract tumors, stricture caused by radiotherapy for colon or cervical cancer, ureteral fistula

Exclusion Criteria:

1. Combine with hypertonic neurogenic bladder (except for patients with long-term indwelling catheter)
2. Colon resection surgery patients -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from ureteral obstruction that require treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Patency rate | Up to 36 months
  Number of patients evaluated with hydronephrosis
Indwelling time | Up to 36 months
  Number of months of the implant in the ureter
Device related serious adverse events | Up to 36 months
  Number of device related serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Peiking university people's hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No